CLINICAL TRIAL: NCT03190785
Title: Benzoic Acid in Beverages: Establishing a Link Between Urinary Metabolites, Metabolic Dysregulation and Weight Loss Failure
Brief Title: Benzoates - an Obesogenic Endocrine Disrupting Chemical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, David Nash Collier, Associate Professor of Pediatrics, East Carolina University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-000376
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: benzoic acid; endocrine disrupting chemicals; leptin; metabolic rate
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Pre/post exposure comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Benzoic acid washout and exposure (Experimental): All subjects will be in this arm which employs a pre-post exposure design. Subjects will undergo a 2 week washout period where they avoid consumption of benzoate containing beverages. Then there is a 1 week exposure period comprising daily consumption of benzoate containing beverages to result in up to 5 mg/kg per day benzoic acid intake.
  Interventions: Other: Benzoic acid washout and exposure

INTERVENTIONS:
Other: Benzoic acid washout and exposure — see above

SUMMARY:
The benzoic acid derivatives sodium and potassium benzoate are preservatives that are commonly added to food and beverages to inhibit microbial growth and prevent spoilage. In the US the major source of benzoate intake is beverages. Studies have shown that piglets or chicks fed low levels of benzoic acid have greater feed efficiency and gain more weight than control fed animals. It has also been shown that benzoic acid inhibits the release of a key metabolic hormone, leptin, from isolated adipocytes (fat cells). Inadequate leptin levels result in increased appetite, decreased metabolic rate, weight gain, insulin resistance and increased diabetes risk.

The primary aim of the proposed research is to directly determine if benzoate consumption in human volunteers results in lower levels of leptin, decreased metabolic rate and increased insulin resistance. If so this would implicate benzoic acid as an obesogen and would help inform more effective approaches to obesity prevention and treatment. A secondary aim of the study is to establish a connection between benzoate exposure and biomarkers in urine that can be used to help treat obese patients.

DETAILED DESCRIPTION:
Our hypothesis is that benzoic acid is an obesogenic xenobiotic that attenuates the leptin signaling pathway resulting in lower metabolic rate and hence a propensity to weight loss non-responsiveness.

This hypothesis will be addressed in this pilot project via the following Specific Aims:

Aim 1. Determine if dietary benzoate attenuates leptin levels and metabolic rate in human subjects. Twenty heathy adolescents and young adults (age 18-25 yrs.) who are either overweight (BMI 25-29.9) or obese (BMI ≥ 30) will be studied. Following a 14 day period of avoiding benzoate containing beverages (washout period) subjects will then consume 36 oz./day of benzoate containing beverages (~ 3.9 - 4.5 mg benzoate/kg body weight per day exposure) for 7 days (exposure period). Fasting plasma samples will be collected pre and post-exposure and leptin, adiponectin, insulin and glucose levels will be compared. Indirect calorimetry will be used to compare resting energy expenditure pre-and post-exposure.

Aim 2. Validate the use of urinary hippurate and glycine to assess benzoate exposure. An early morning void urine samples will be collected pre-and post-exposure. Non-targeted NMR-based metabolomics analysis will be used to compare changes in individual subject's urinary metabolome using pre- and post-exposure as the "phenotypic" anchors.

ELIGIBILITY:
Inclusion Criteria:

* Young adult (18-30 yrs)
* Healthy non-smoker
* Either overweight (BMI >25 but <30) or obese (BMI >30)
* Has or can obtain transportation to study site
* Able to provide written consent in English

Exclusion Criteria:

* Metabolic disease

  1. Diabetes mellitus
  2. Hypothyroidism
* Use of medication that may influence metabolism

  1. Anti-hyperglycemic agents
  2. Thyroid hormone
  3. Stimulants for ADD/ADHD
  4. Atypical anti-psychotics
  5. Weight loss medications
* Benzoate sensitivity
* Known pregnancy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Metabolic rate | measured following 1 week dietary exposure to benzoic acid.
  Metabolic rate as measured by indirect calorimetry

SECONDARY OUTCOMES:
Leptin levels | measured following 1 week dietary exposure to benzoic acid
  Circulating levels of the adipokine leptin will be measured using ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Brody School of Medicine at East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No